CLINICAL TRIAL: NCT02966613
Title: Primary TKA Using a Fully Disposable Patient-Specific Instrumentation: A Multicenter Controlled Study
Brief Title: Fully Disposable Patient-Specific Instrumentation
Acronym: MyKnee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochin Hospital (Ambiguous)
Responsible Party: Principal Investigator, Moussa Hamadouche, MD, PhD, Professor of Orthopaedic Surgery, Cochin Hospital
Organization: Cochin Hospital, India (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SC2900
Record Dates: First submitted 2016-09-26; First posted 2016-11-17 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Osteoarthritis,Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CI (Active Comparator): TKA using conventional instrumentation (CI)
  Interventions: Device: GMK Medacta Total Knee arthroplasty
- PSCG (Experimental): TKA performed using Patient specific cutting guides (PSCG)
  Interventions: Device: GMK Medacta Total Knee arthroplasty
- PSCG-D (Experimental): TKA performed using fully disposable Patient specific cutting guides (PSCG-D)
  Interventions: Device: GMK Medacta Total Knee arthroplasty

INTERVENTIONS:
Device: GMK Medacta Total Knee arthroplasty — Total Knee arthroplasty

SUMMARY:
To evaluate the lower limb alignment following total knee arthroplasty (TKA) performed with fully disposable patient-specific instrumentation versus conventional, versus patient specific instrumentation.

DETAILED DESCRIPTION:
The investigators performed a controlled multicenter trial comparing the clinical and radiologic results and resources consumption of primary TKA using patient-specific cutting guides (PSCG) versus conventional instrumentation (CI), and compared the results to those obtained with a fully disposable patient-specific instrumentation (PSCG-D).

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 18 and 85 years
* able to understand information
* affiliated to social security

Exclusion Criteria:

* active or suspected sepsis
* tumor around the knee
* previous partial or total knee replacement
* extra-articular deformation requiring osteotomy around the knee in conjunction with TKA
* social situation that could impair follow-up

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
HKA angle | 3 months
  Lower limb mechanical axis was measured on a bipodal standing leg-length anteroposterior radiograph with the patella oriented straight made three months postoperatively, using Roman software version 1.70 (Oswestry, United Kingdom). Postoperative lower limb mechanical axis was calculated from the Hip-Knee-Ankle (HKA) angle between the femoral and tibial mechanical axes, respectively. An HKA angle greater than 180° was indicative of valgus, whereas values lower than 180° indicated varus.

SECONDARY OUTCOMES:
% outliers | 3 months
  % of patients with an HKA angle outside 180°+/- 3°
Knee Society Score | 3 months
  Validated pain and function score following TKA
Oxford Knee Score | 3 months
  Patients self assessment of knee function

REFERENCES:
- [Derived] Abane L, Zaoui A, Anract P, Lefevre N, Herman S, Hamadouche M. Can a Single-Use and Patient-Specific Instrumentation Be Reliably Used in Primary Total Knee Arthroplasty? A Multicenter Controlled Study. J Arthroplasty. 2018 Jul;33(7):2111-2118. doi: 10.1016/j.arth.2018.02.038. Epub 2018 Feb 17. PMID 29576488